CLINICAL TRIAL: NCT02883231
Title: Plasma Level of Mitochondrial DNA in Patients With ARDS and Its Clinical Significance
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Chun Pan (Other)
Responsible Party: Sponsor-Investigator, Chun Pan, attending doctor, Southeast University, China
Organization: Southeast University, China (Other)
Other Study IDs: ARDS mtDNA
Record Dates: First submitted 2016-08-25; First posted 2016-08-30 (Estimated); Last update posted 2016-08-30 (Estimated); Status verified 2016-08

CONDITIONS: Evaluate the Correlation Between the Level of Mitochondrial DNA in Plasma and the Prognosis of the Patients With ARDS.

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: taking peripheral blood — taking peripheral blood of no more than 3ml

SUMMARY:
To observe the changes of plasma mitochondrial DNA (mtDNA) levels in patients with ARDS, and to explore its clinical significance.

DETAILED DESCRIPTION:
60 patients who diagnosed as ARDS were included in this study.Then keep blood samples from these patients in the first day、the third day and the sveventh day,detect the mitochotndrial DNA level in plasma by real-time quantitative PCR. Recored Severity of illness and survival status of every patient within 28 days.Objective to evaluate the correlation between the level of mitochondrial DNA in plasma and the prognosis of the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients admitted to ICU diagnosed of ARDS (Berlin criteria),
2. Patients age between 18 years old and 80 years.

Exclusion Criteria:

1. Pregnant women,
2. Patients with malignant tumor,
3. Immunosuppression or immunocompromised patients.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population admitted to ICU of Zhongda hospital ，diagnosed of ARDS。
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-04; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
mortality | 28-day

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Peng F, Liang C, Chang W, Sun Q, Xie J, Qiu H, Yang Y. Prognostic Significance of Plasma Hepatocyte Growth Factor in Sepsis. J Intensive Care Med. 2022 Mar;37(3):352-358. doi: 10.1177/0885066621993423. Epub 2021 Feb 22. PMID 33611982